CLINICAL TRIAL: NCT06230575
Title: Locoregional Blocks for Breast Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Assistant professor of Anesthesia, Surgical Critical care and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AP2312-301-072
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- erector spinae block (Active Comparator): Erector spinae plane block on the ipsilateral operative site
  Interventions: Procedure: erector spinae block
- retrolaminar block (Experimental): Retrolaminar plane block on the ipsilateral operative site
  Interventions: Procedure: retrolaminar block
- serratus anterior block (Experimental): Serratus anterior plane block on the ipsilateral operative site
  Interventions: Procedure: serratus anterior block
- pectoral nerve block II (Experimental): Pectoral nerve block II on the ipsilateral operative site
  Interventions: Procedure: pectoral nerve block

INTERVENTIONS:
Procedure: erector spinae block — Erector spinae plane block
  Arms: erector spinae block
Procedure: retrolaminar block — Retrolaminar block
  Arms: retrolaminar block
Procedure: serratus anterior block — Serratus anterior plane block
  Arms: serratus anterior block
Procedure: pectoral nerve block — Pectoral nerve block
  Arms: pectoral nerve block II

SUMMARY:
Breast surgeries are common operative procedures that require appropriate postoperative analgesia.

DETAILED DESCRIPTION:
Numerous pain relief techniques, including several new regional anesthesia techniques, are available for control of acute pain after breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* female cancer breast patient
* age from 18- 65

Exclusion Criteria:

* coagulation defect
* Patient refusal
* abnormal kidney and or liver function tests

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with breast cancer
Enrollment: 188 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
time to receive first postoperative analgesic | First 24 hours postoperatively
  time to first dose of rescue opioid analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Assistant professor of Anesthesia, Surgical critical care and Pain Management, National Cancer Institute, Cairo University
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt